CLINICAL TRIAL: NCT04480021
Title: Mobile Mental Health in Community-Based Organizations: A Stepped Care Approach to Women's Mental Health
Brief Title: Mobile Mental Health in Community-Based Organizations
Acronym: MITHRA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Amritha Subray Bhat, Assistant Professor, Psychiatry, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: STUDY00010415; R21MH124073-01 (NIH)
Record Dates: First submitted 2020-07-10; First posted 2020-07-21 (Actual); Results first posted 2024-08-13 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-07

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multiuser Interactive Health Response Application (MITHRA) (Experimental): Randomization is at the level of the Community Based Organization (CBO). CBOs randomized to MITHRA will have access to the MITHRA app on tablets. MITHRA app will include depression screening and behavioral activation modules.
  Interventions: Behavioral: MITHRA
- Enhanced Usual Care (EUC) (Placebo Comparator): CBOs randomized to EUC will receive standardized monthly group education (45 min) regarding the symptoms of depression
  Interventions: Behavioral: EUC

INTERVENTIONS:
Behavioral: MITHRA — A mobile based application (app) in CBOs to screen, track and treat mild to moderate depression among low income women using Healthy Activity Program (HAP),a WHO-recommended evidence-based intervention.
  Arms: Multiuser Interactive Health Response Application (MITHRA)
Behavioral: EUC — Group education on depression by community health workers
  Arms: Enhanced Usual Care (EUC)

SUMMARY:
Untreated depression is a significant cause of morbidity and mortality among women in low and middle- income countries (LMIC). The investigators propose to develop and test the feasibility an interactive voice-response, mobile health application (MITHRA) for screening, tracking symptom severity and supporting stepped treatment of depression among women in rural India. The study will lead to the development of a scalable mobile application applicable to other low resource settings, and build research capacity at the India site.

DETAILED DESCRIPTION:
Undiagnosed and untreated depression is a significant cause of morbidity and mortality in low-, middle-income countries (LMIC) such as India. The rates of diagnosis and treatment of depression among women in rural India are disproportionately low despite a primary care based task-sharing model of mentalhealth treatment. Stepped care approaches support appropriate treatment of symptoms while reducing the burden on healthcare systems and mobile technology can reduce the mental health treatment gap given its reach and easy access. However, our preliminary study at a task-sharing care model in rural south India revealed that illiteracy and the practice of sharing mobile phones as a family resource present hurdles to the adoption of mobile mental health (mHealth) based interventions. To date, the feasibility of a community based multiple user mHealth application to screen depression, track symptom severity and support the delivery of stepped care treatment has not been tested in LMIC.

Specific Aim 1: In phase I of this exploratory study, the investigators will adopt a user centered participatory approach to design and develop a multiple-user, voice-response, mobile application ("MITHRA"), to be used in community-based organizations for screening, tracking and supporting stepped care treatment for depression, including select modules of the Healthy Activity Program, a brief psychological intervention based on behavioral activation. The application will include audio, video and enhanced touchscreen capabilities, to overcome the barrier of illiteracy and lack of access.

Specific Aim 2: In phase II, using a randomized-control design, the investigators will examine feasibility and utility of "MITHRA" deployed at community-based organizations (n=3) vs enhanced usual care (n=3) in community-based organizations (enrolling approximately 60 women).

Specific aim 3: Throughout the duration of the funding period the investigators will arrange for mentored participation of Psychiatry and Community Medicine residents from India in the research project with involvement in the entire spectrum of research activities from interview development and conduct to qualitative and quantitative data analysis and manuscript writing and dissemination. This mentored participation will be supported by regular video-conferenced didactic and case presentation sessions on research methodology.

The grant will accomplish the goals of developing a unique mobile application that is scalable, examining its feasibility and building research capacity at the research site in India.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Resident of the village (i.e. not a guest attendee)
* Plans to attend CBO meetings regularly.

Exclusion Criteria:

* Diagnosed with severe mental illness such as bipolar disorder or schizophrenia (measured by self report / socio demographic questionnaire)
* Suicide attempt or severe alcohol or substance use in the past 6 months (measured by self report / socio demographic questionnaire)
* Unable to participate in informed consent discussion

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Enrollment: 85 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-08-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amritha S Bhat, MD, MPH, Principal Investigator — University of Washington
Locations (1):
- St. John's Research Institute, Bengaluru, India

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Multiuser Interactive Health Response Application (MITHRA) | Enhanced Usual Care (EUC)
Started | 49 | 36
Completed | 46 | 32
Not Completed | 3 | 4
Not completed — Lost to Follow-up | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Multiuser Interactive Health Response Application (MITHRA) | Enhanced Usual Care (EUC) | Total
Number analyzed (Participants) | 49 | 36 | 85
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.6 (10.5) | 40.7 (11.9) | 41.2 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 36 | 85
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 49 | 36 | 85
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 49 | 36 | 85
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  India | 49 | 36 | 85
QIDS-SR [Median (Inter-Quartile Range); unit: units on a scale] — Quick Inventory of Depressive Symptomatology Range of scores 0 to 27 with higher scores indicating more depressive symptoms
  units on a scale | 4.0 [2.0 to 5.0] | 2.5 [0 to 4.0] | 3.0 [2.0 to 5.0]

OUTCOME MEASURES:

1. Primary Outcome: Usage Rates
Description: The investigators will obtain data on women's rates of use of the MITHRA app - this data will be obtained from the app, enabled by the single user sign on. Only the MITHRA arm will be considered, and completion of 50% of modules will be considered adequate usage.
Time Frame: 3 months
Population: Usage rates only calculated for those assigned to intervention.
Measure: Number; unit: participants
Arm/Group | Multiuser Interactive Health Response Application (MITHRA)
Number analyzed (Participants) | 49
participants | 47

2. Secondary Outcome: Depression
Description: Change in Quick Inventory of Depressive Symptomatology Self Report (QIDS SR - a self report tool used to measure symptoms of depression) which will be collected by a blinded / masked research assistant. Research assessments will be conducted over the phone or in the Primary Health Center to avoid unblinding of CBO randomization status (presence of tablets in the CBOs) Scores range from 0 to 27 with higher scores indicating more symptoms
Time Frame: Change from baseline depression score (QIDS SR) at 3 months
Population: Participants with assessments available at 3 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Multiuser Interactive Health Response Application (MITHRA) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 47 | 31
score on a scale | 0 [-2.0 to 1.0] | 0 [-2.0 to 1.0]

3. Secondary Outcome: Depression
Description: Change in Quick Inventory of Depressive Symptomatology Self Report (QIDS SR - a self report tool used to measure symptoms of depression) which will be collected by a blinded / masked research assistant. Research assessments will be conducted over the phone or in the Primary Health Center to avoid unblinding of CBO randomization status (presence of tablets in the CBOs) Range of scores is 0 to 27, with higher scores indicated more symptoms
Time Frame: Change from baseline depression score (QIDS SR) at 6 months
Population: Participants with assessments available at 6 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Multiuser Interactive Health Response Application (MITHRA) | Enhanced Usual Care (EUC)
Number analyzed (Participants) | 46 | 32
score on a scale | -1.0 [-3.0 to 1.0] | 0 [-0.75 to 2.75]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Multiuser Interactive Health Response Application (MITHRA) | Enhanced Usual Care (EUC)
All-Cause Mortality (participants affected / at risk) | 0/49 | 0/36
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/36
Other Adverse Events (participants affected / at risk) | 0/49 | 0/36

LIMITATIONS AND CAVEATS:
Women with severe depression may not attend Self Help Group meetings. The intervention would ideally include a way to involve women with severe depressive symptoms, and ensure that they get the appropriate level of care.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-07-16): https://cdn.clinicaltrials.gov/large-docs/21/NCT04480021/Prot_SAP_ICF_000.pdf